CLINICAL TRIAL: NCT02211261
Title: A Phase 1 Double-blind, Placebo-controlled, Randomized, Single- And Multiple-ascending Dose Study To Assess The Safety, Tolerability, And Pharmacokinetics Of Pf-06293620 In Subjects With Type 2 Diabetes Mellitus
Brief Title: A Phase 1 Single/Multiple Dose Study Of PF-06293620 To Assess Safety, Tolerability And Pharmacokinetics In Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B3501001
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: first in human; single dose; multiple dose; escalation; safety study; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — RN909

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Cohort 1-PF-06293620 or placebo (Experimental): Single Ascending Dose PF-06293620 or placebo
  Interventions: Biological: PF-06293620; Biological: Placebo
- Cohort 2-PF-06293620 or placebo (Experimental): Single Ascending Dose PF-06293620 or placebo
  Interventions: Biological: PF-06293620; Biological: Placebo
- Cohort 3-PF-06293620 or placebo (Experimental): Single Ascending Dose PF-06293620 or placebo
  Interventions: Biological: PF-06293620; Biological: Placebo
- Cohort 4-PF-06293620 or placebo (Experimental): Single Ascending Dose PF-06293620 or placebo
  Interventions: Biological: PF-06293620; Biological: Placebo
- Cohort 5-PF-06293620 or placebo (Experimental): Single Ascending Dose PF-06293620 or placebo
  Interventions: Biological: PF-06293620; Biological: Placebo
- Cohort 6-PF-06293620 or placebo (Experimental): Multiple Ascending Dose PF-06293620 or placebo
  Interventions: Biological: PF-06293620; Biological: Placebo
- Cohort 7 PF-06293620 or placebo (Experimental): Multiple Ascending Dose PF-06293620 or placebo
  Interventions: Biological: PF-06293620; Biological: Placebo
- Cohort 8-PF-06293620 or placebo (Experimental): Multiple Ascending Dose PF-06293620 or placebo
  Interventions: Biological: PF-06293620; Biological: Placebo
- Cohort 9-PF-06293620 or placebo (Experimental): Multiple Ascending Dose PF-06293620 or placebo
  Interventions: Biological: PF-06293620; Biological: Placebo

INTERVENTIONS:
Biological: PF-06293620 — subcutaneous, single dose 0.3 mg/kg
  Arms: Cohort 1-PF-06293620 or placebo
Biological: Placebo — Subcutaneous normal saline single dose
  Arms: Cohort 1-PF-06293620 or placebo
Biological: PF-06293620 — Subcutaneous, single dose 1.0 mg/kg
  Arms: Cohort 2-PF-06293620 or placebo
Biological: Placebo — Subcutaneous normal saline single dose
  Arms: Cohort 2-PF-06293620 or placebo
Biological: PF-06293620 — Subcutaneous single dose 3 mg/kg
  Arms: Cohort 3-PF-06293620 or placebo
Biological: Placebo — Subcutaneous normal saline single dose
  Arms: Cohort 3-PF-06293620 or placebo
Biological: PF-06293620 — Subcutaneous single dose 6 mg/kg
  Arms: Cohort 4-PF-06293620 or placebo
Biological: Placebo — Subcutaneous normal saline single dose
  Arms: Cohort 4-PF-06293620 or placebo
Biological: PF-06293620 — Intravenous infusion single dose 1 mg/kg
  Arms: Cohort 5-PF-06293620 or placebo
Biological: Placebo — Intravenous infusion normal saline single dose
  Arms: Cohort 5-PF-06293620 or placebo
Biological: PF-06293620 — Subcutaneous injection multiple dose 75 mg (Days 1, 29 and 57)
  Arms: Cohort 6-PF-06293620 or placebo
Biological: Placebo — Subcutaneous injection normal saline multiple dose (Days 1, 29 and 57)
  Arms: Cohort 6-PF-06293620 or placebo
Biological: PF-06293620 — Subcutaneous injection multiple dose 150 mg (Days 1, 29 and 57)
  Arms: Cohort 7 PF-06293620 or placebo
Biological: Placebo — Subcutaneous injection normal saline multiple dose (Days 1, 29 and 57)
  Arms: Cohort 7 PF-06293620 or placebo
Biological: PF-06293620 — Subcutaneous injection multiple dose 250 mg (Days 1, 29 and 57)
  Arms: Cohort 8-PF-06293620 or placebo
Biological: Placebo — Subcutaneous injection normal saline multiple dose (Days 1, 29 and 57)
  Arms: Cohort 8-PF-06293620 or placebo
Biological: PF-06293620 — Subcutaneous injection multiple dose TBD mg (Days TBD)
  Arms: Cohort 9-PF-06293620 or placebo
Biological: Placebo — Subcutaneous injection normal saline multiple dose (Days TBD)
  Arms: Cohort 9-PF-06293620 or placebo

SUMMARY:
A first in human study to determine the safety, tolerability and pharmacokinetics of single and multiple ascending doses of PF-06293620 in subjects with Type 2 Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria:

* Men and women of non-childbearing potential with Type 2 Diabetes Mellitus
* Subjects on stable doses of metformin >/= 1500 mg daily (SAD cohorts) or >/= 1000 mg daily (MAD cohorts) x 30 days prior to screening
* HbA1c 7-10% (SAD Cohorts) or 6.5-10% (MAD cohorts) inclusive at screening
* Fasting C-peptide >1.12 ng/mL (SAD cohorts) or >/= 0.8 mg/mL (MAD cohorts) at screening

Exclusion Criteria:

* History of Type 1 diabetes mellitus
* Evidence of diabetic complications with significant end-organ damage
* History of chronic pancreatitis or at high risk for pancreatitis
* Poorly controlled hypertension
* History of cardiovascular or cerebrovascular event or procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-09-15 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Profil Institute for Clinical Research, Inc., Chula Vista, California
  - Profil Institute for Clinical Research, Incorporated, Chula Vista, California
  - Avail Clinical Research, LLC, DeLand, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Qps Mra, Llc, South Miami, Florida
  - Qps-Mra Llc, South Miami, Florida
  - High Point Clinical Trials Center, LLC, High Point, North Carolina

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3501001&StudyName=A%20Phase%201%20Single%20Dose%20Study%20Of%20PF-06293620%20To%20Assess%20Safety%2C%20Tolerability%20And%20Pharmacokinetics%20In%20Subjects%20With%20Type%202%20Diabetes%20Mell

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo SC (SAD Cohorts): One group of participants in the single-ascending dose (SAD) cohorts received a single dose of placebo matched to PF-06293620 by subcutaneous (SC) injection to the abdomen following an overnight fast of at least 10 hours.
- PF-06293620 0.3 mg/kg SC (SAD Cohorts): One group of participants in the single-ascending dose (SAD) cohorts received a single dose of PF-06293620 at 0.3 mg/kg by subcutaneous (SC) injection to the abdomen following an overnight fast of at least 10 hours.
- PF-06293620 1.0 mg/kg SC (SAD Cohorts): One group of participants in the single-ascending dose (SAD) cohorts received a single dose of PF-06293620 at 1.0 mg/kg by subcutaneous (SC) injection to the abdomen following an overnight fast of at least 10 hours.
- PF-06293620 3.0 mg/kg SC (SAD Cohorts): One group of participants in the single-ascending dose (SAD) cohorts received a single dose of PF-06293620 at 3.0 mg/kg by subcutaneous (SC) injection to the abdomen following an overnight fast of at least 10 hours.
- PF-06293620 6.0 mg/kg SC (SAD Cohorts): One group of participants in the single-ascending dose (SAD) cohorts received a single dose of PF-06293620 at 6.0 mg/kg by subcutaneous (SC) injection to the abdomen following an overnight fast of at least 10 hours.
- Placebo IV (SAD Cohorts): One group of participants in the single-ascending dose (SAD) cohorts received a single dose of placebo matched to PF-06293620 by intravenous (IV) infusion over approximately 60 minutes following an overnight fast of at least 10 hours.
- PF-06293620 1.0 mg/kg IV (SAD Cohorts): One group of participants in the single-ascending dose (SAD) cohorts received a single dose of PF-06293620 at 1.0 mg/kg by intravenous (IV) infusion over approximately 60 minutes following an overnight fast of at least 10 hours.
- Placebo SC (MAD Cohorts): One group of participants in the multiple-ascending dose (MAD) cohorts received placebo matched to PF-06293620 every 4 weeks (on Days 1, 29 and 57, deviation of plus or minus 2 days was allowed for Day 29 and Day 57 dosing) by subcutaneous (SC) injection to the abdomen following an overnight fast of at least 10 hours.
- PF-06293620 50 mg SC (MAD Cohorts): One group of participants in the multiple-ascending dose (MAD) cohorts received PF-06293620 50 mg every 4 weeks (on Days 1, 29 and 57, deviation of plus or minus 2 days was allowed for Day 29 and Day 57 dosing) by subcutaneous (SC) injection to the abdomen following an overnight fast of at least 10 hours.
- PF-06293620 75 mg SC (MAD Cohorts): One group of participants in the multiple-ascending dose (MAD) cohorts received PF-06293620 75 mg every 4 weeks (on Days 1, 29 and 57, deviation of plus or minus 2 days was allowed for Day 29 and Day 57 dosing) by subcutaneous (SC) injection to the abdomen following an overnight fast of at least 10 hours.
- PF-06293620 150 mg SC (MAD Cohorts): One group of participants in the multiple-ascending dose (MAD) cohorts received PF-06293620 150 mg every 4 weeks (on Days 1, 29 and 57, deviation of plus or minus 2 days was allowed for Day 29 and Day 57 dosing) by subcutaneous (SC) injection to the abdomen following an overnight fast of at least 10 hours.
Period: Overall Study
Arm/Group | Placebo SC (SAD Cohorts) | PF-06293620 0.3 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg SC (SAD Cohorts) | PF-06293620 3.0 mg/kg SC (SAD Cohorts) | PF-06293620 6.0 mg/kg SC (SAD Cohorts) | Placebo IV (SAD Cohorts) | PF-06293620 1.0 mg/kg IV (SAD Cohorts) | Placebo SC (MAD Cohorts) | PF-06293620 50 mg SC (MAD Cohorts) | PF-06293620 75 mg SC (MAD Cohorts) | PF-06293620 150 mg SC (MAD Cohorts)
Started | 9 | 6 | 6 | 6 | 9 | 2 | 6 | 8 | 8 | 16 | 8
Completed | 9 | 6 | 5 | 6 | 7 | 1 | 6 | 7 | 8 | 14 | 8
Not Completed | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo SC (SAD Cohorts) | PF-06293620 0.3 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg SC (SAD Cohorts) | PF-06293620 3.0 mg/kg SC (SAD Cohorts) | PF-06293620 6.0 mg/kg SC (SAD Cohorts) | Placebo IV (SAD Cohorts) | PF-06293620 1.0 mg/kg IV (SAD Cohorts) | Placebo SC (MAD Cohorts) | PF-06293620 50 mg SC (MAD Cohorts) | PF-06293620 75 mg SC (MAD Cohorts) | PF-06293620 150 mg SC (MAD Cohorts) | Total
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 9 | 2 | 6 | 8 | 8 | 16 | 8 | 84
Age, Customized [Number; unit: participants]
  <18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18-44 years | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3
  45-64 years | 7 | 4 | 4 | 6 | 6 | 1 | 5 | 7 | 4 | 9 | 8 | 61
  >=65 years | 2 | 2 | 2 | 0 | 2 | 0 | 0 | 1 | 4 | 7 | 0 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 4 | 3 | 4 | 0 | 0 | 4 | 3 | 9 | 1 | 34
  Male | 4 | 5 | 2 | 3 | 5 | 2 | 6 | 4 | 5 | 7 | 7 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 2 | 4 | 3 | 2 | 4 | 2 | 4 | 7 | 7 | 46
  Not Hispanic or Latino | 3 | 1 | 4 | 2 | 6 | 0 | 2 | 6 | 4 | 9 | 1 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-Causality and Treatment Related Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device, regardless of its causal relationship with study treatment. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; was life-threatening (immediate risk of death); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs are events between first dose of study drug and up to Day 85 (for SAD cohorts) or Day 169 (for MAD cohorts) that were absent before treatment or that worsened after treatment. AEs included both serious and non-serious AEs. Causality with the study treatment was determined by the investigator.
Time Frame: Days 1 to 85 for SAD cohorts and Days 1 to 169 for MAD cohorts; participants with positive anti-drug antibody (ADA) results were followed up to stabilization of ADA titers or up to 9 months after Day 169 visit.
Population: The safety analysis population included all participants who received any amount of dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo SC (SAD Cohorts) | PF-06293620 0.3 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg SC (SAD Cohorts) | PF-06293620 3.0 mg/kg SC (SAD Cohorts) | PF-06293620 6.0 mg/kg SC (SAD Cohorts) | Placebo IV (SAD Cohorts) | PF-06293620 1.0 mg/kg IV (SAD Cohorts) | Placebo SC (MAD Cohorts) | PF-06293620 50 mg SC (MAD Cohorts) | PF-06293620 75 mg SC (MAD Cohorts) | PF-06293620 150 mg SC (MAD Cohorts)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 9 | 2 | 6 | 8 | 8 | 16 | 8
participants
  All-causality AE | 5 | 3 | 3 | 5 | 5 | 0 | 3 | 4 | 4 | 11 | 8
  All-causality SAE | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Treatment-related AE | 1 | 0 | 0 | 3 | 3 | 0 | 1 | 1 | 1 | 4 | 5
  Treatment-related SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Dose Limiting or Intolerable Adverse Events
Description: Dose limiting or intolerable AEs were originally planned to be collected. However, this outcome measure was not actually summarized, since collection and monitoring of treatment-emergent AEs was performed during the study, and deemed sufficient to ensure the participants safety.
Time Frame: Days 1 to 85 for SAD cohorts; Days 1 to 169 for MAD Cohorts
Population: Data for this outcome measure were not collected.
Arm/Group | Placebo SC (SAD Cohorts) | PF-06293620 0.3 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg SC (SAD Cohorts) | PF-06293620 3.0 mg/kg SC (SAD Cohorts) | PF-06293620 6.0 mg/kg SC (SAD Cohorts) | Placebo IV (SAD Cohorts) | PF-06293620 1.0 mg/kg IV (SAD Cohorts) | Placebo SC (MAD Cohorts) | PF-06293620 50 mg SC (MAD Cohorts) | PF-06293620 75 mg SC (MAD Cohorts) | PF-06293620 150 mg SC (MAD Cohorts)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Positive Anti-drug Antibody (ADA) Result
Description: ADA against PF-06293620 in human serum samples was determined following a tiered approach using screening, confirmation, and titer/quantification by semi-quantitative enzyme linked immunosorbent assay (ELISA). Endpoint titer >=1.88 was considered positive.
Time Frame: Days 1 to 85 for SAD cohorts; Days 1 to 169 for MAD Cohorts
Population: The safety analysis population included all participants who received any amount of dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo SC (SAD Cohorts) | PF-06293620 0.3 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg SC (SAD Cohorts) | PF-06293620 3.0 mg/kg SC (SAD Cohorts) | PF-06293620 6.0 mg/kg SC (SAD Cohorts) | Placebo IV (SAD Cohorts) | PF-06293620 1.0 mg/kg IV (SAD Cohorts) | Placebo SC (MAD Cohorts) | PF-06293620 50 mg SC (MAD Cohorts) | PF-06293620 75 mg SC (MAD Cohorts) | PF-06293620 150 mg SC (MAD Cohorts)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 9 | 2 | 6 | 8 | 8 | 16 | 8
participants | 1 | 5 | 2 | 1 | 2 | 0 | 1 | 0 | 5 | 7 | 4

4. Secondary Outcome: Area Under the Serum Concentration-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of PF-06293620 (SAD Cohorts)
Description: AUCinf was calculated as AUClast +(Clast*/kel), where AUClast is area under the serum concentration-time profile from time 0 to the time of the last quantifiable concentration, Clast* is the predicted serum concentration at the last quantifiable time point estimated from the log-linear regression analysis, kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Only those data points judged to describe the terminal log-linear decline were used in the regression.
Time Frame: Pre-dose, 1, 4, 8 and 12 hours post-dose on Day 1; 24 and 36 hours post-dose on Day 2; Days 3, 4, 5, 8, 15, 22, 29, 43, 57, 85
Population: The PK parameter analysis population included all participants randomized and treated who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/milliliter (mcg*hr/mL)
Arm/Group | PF-06293620 0.3 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg SC (SAD Cohorts) | PF-06293620 3.0 mg/kg SC (SAD Cohorts) | PF-06293620 6.0 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg IV (SAD Cohorts)
Number analyzed (Participants) | 1 | 5 | 6 | 7 | 6
microgram*hour/milliliter (mcg*hr/mL) | 300 (NA) — Only 1 participant had reportable value, geometric coefficient of variation is not applicable. | 1716 (46) | 6306 (54) | 19440 (56) | 6775 (12)

5. Secondary Outcome: Dose-normalized AUCinf (AUCinf(dn)) of PF-06293620 (SAD Cohorts)
Description: AUCinf(dn) was calculated as AUCinf/dose, where AUCinf is area under the serum concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL/mg
Arm/Group | PF-06293620 0.3 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg SC (SAD Cohorts) | PF-06293620 3.0 mg/kg SC (SAD Cohorts) | PF-06293620 6.0 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg IV (SAD Cohorts)
Number analyzed (Participants) | 1 | 5 | 6 | 7 | 6
mcg*hr/mL/mg | 12.00 (NA) — Only 1 participant had reportable value, geometric coefficient of variation is not applicable. | 22.24 (45) | 23.79 (47) | 36.13 (49) | 67.94 (16)
Statistical Analysis 1: Comparison: PF-06293620 0.3 mg/kg SC (SAD Cohorts) vs PF-06293620 1.0 mg/kg IV (SAD Cohorts); Test type: Other; Percentage of Test relative to Reference = 17.66, 90% CI 2-sided [8.44 to 36.95] — PF-06293620 0.3 mg/kg SC (SAD Cohorts) is Test, PF-06293620 1.0 mg/kg IV (SAD Cohorts) is Reference
Statistical Analysis 2: Comparison: PF-06293620 1.0 mg/kg SC (SAD Cohorts) vs PF-06293620 1.0 mg/kg IV (SAD Cohorts); Test type: Other; Percentage of Test relative to Reference = 32.73, 90% CI 2-sided [21.64 to 49.51] — PF-06293620 1.0 mg/kg SC (SAD Cohorts) is Test, PF-06293620 1.0 mg/kg IV (SAD Cohorts) is Reference
Statistical Analysis 3: Comparison: PF-06293620 3.0 mg/kg SC (SAD Cohorts) vs PF-06293620 1.0 mg/kg IV (SAD Cohorts); Test type: Other; Percentage of Test relative to Reference = 35.02, 90% CI 2-sided [23.60 to 51.95] — PF-06293620 3.0 mg/kg SC (SAD Cohorts) is Test, PF-06293620 1.0 mg/kg IV (SAD Cohorts) is Reference
Statistical Analysis 4: Comparison: PF-06293620 6.0 mg/kg SC (SAD Cohorts) vs PF-06293620 1.0 mg/kg IV (SAD Cohorts); Test type: Other; Percentage of Test relative to Reference = 53.18, 90% CI 2-sided [36.36 to 77.78] — PF-06293620 6.0 mg/kg SC (SAD Cohorts) is Test, PF-06293620 1.0 mg/kg IV (SAD Cohorts) is Reference

6. Secondary Outcome: Area Under the Serum Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of PF-06293620 (SAD Cohorts)
Description: Area under the serum concentration-time profile from time 0 to the time of the last quantifiable concentration (AUClast) of PF-06293620 was determined using linear/log trapezoidal method.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL
Arm/Group | PF-06293620 0.3 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg SC (SAD Cohorts) | PF-06293620 3.0 mg/kg SC (SAD Cohorts) | PF-06293620 6.0 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg IV (SAD Cohorts)
Number analyzed (Participants) | 5 | 5 | 6 | 7 | 6
mcg*hr/mL | 128.3 (54) | 1619 (46) | 5945 (53) | 18080 (58) | 6509 (13)

7. Secondary Outcome: Dose-normalized AUClast (AUClast(dn)) of PF-06293620 (SAD Cohorts)
Description: AUClast(dn) of PF-06293620 was calculated as AUClast/dose, where AUClast was area under the serum concentration-time profile from time 0 to the time of the last quantifiable concentration.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL/mg
Arm/Group | PF-06293620 0.3 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg SC (SAD Cohorts) | PF-06293620 3.0 mg/kg SC (SAD Cohorts) | PF-06293620 6.0 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg IV (SAD Cohorts)
Number analyzed (Participants) | 5 | 5 | 6 | 7 | 6
mcg*hr/mL/mg | 4.779 (58) | 21.01 (44) | 22.47 (47) | 33.59 (50) | 65.26 (18)
Statistical Analysis 1: Comparison: PF-06293620 0.3 mg/kg SC (SAD Cohorts) vs PF-06293620 1.0 mg/kg IV (SAD Cohorts); Test type: Other; Percentage of Test relative to Reference = 7.32, 90% CI 2-sided [4.70 to 11.40] — PF-06293620 0.3 mg/kg SC (SAD Cohorts) is Test, PF-06293620 1.0 mg/kg IV (SAD Cohorts) is Reference
Statistical Analysis 2: Comparison: PF-06293620 1.0 mg/kg SC (SAD Cohorts) vs PF-06293620 1.0 mg/kg IV (SAD Cohorts); Test type: Other; Percentage of Test relative to Reference = 32.19, 90% CI 2-sided [20.67 to 50.12] — PF-06293620 1.0 mg/kg SC (SAD Cohorts) is Test, PF-06293620 1.0 mg/kg IV (SAD Cohorts) is Reference
Statistical Analysis 3: Comparison: PF-06293620 3.0 mg/kg SC (SAD Cohorts) vs PF-06293620 1.0 mg/kg IV (SAD Cohorts); Test type: Other; Percentage of Test relative to Reference = 34.43, 90% CI 2-sided [22.57 to 52.52] — PF-06293620 3.0 mg/kg SC (SAD Cohorts) is Test, PF-06293620 1.0 mg/kg IV (SAD Cohorts) is Reference
Statistical Analysis 4: Comparison: PF-06293620 6.0 mg/kg SC (SAD Cohorts) vs PF-06293620 1.0 mg/kg IV (SAD Cohorts); Test type: Other; Percentage of Test relative to Reference = 51.47, 90% CI 2-sided [34.26 to 77.31] — PF-06293620 6.0 mg/kg SC (SAD Cohorts) is Test, PF-06293620 1.0 mg/kg IV (SAD Cohorts) is Reference

8. Secondary Outcome: Clearance (CL) of PF-06293620 (SAD Cohorts)
Description: Clearance (CL) was calculated as dose/AUCinf, where AUCinf was area under the serum concentration-time profile from time 0 extrapolated to infinite time. This outcome measure only applies to IV arms.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | PF-06293620 1.0 mg/kg IV (SAD Cohorts)
Number analyzed (Participants) | 6
mL/hr | 14.72 (16)

9. Secondary Outcome: Apparent Clearance (CL/F) of PF-06293620 (SAD Cohorts)
Description: Apparent Clearance (CL/F) of PF-06293620 was calculated as dose/AUCinf, where AUCinf was area under the serum concentration-time profile from time 0 extrapolated to infinite time. This outcome measure only applies to SC arms.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | PF-06293620 0.3 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg SC (SAD Cohorts) | PF-06293620 3.0 mg/kg SC (SAD Cohorts) | PF-06293620 6.0 mg/kg SC (SAD Cohorts)
Number analyzed (Participants) | 1 | 5 | 6 | 7
mL/hr | 83.20 (NA) — Only 1 participant had reportable value, geometric coefficient of variation is not applicable. | 44.93 (45) | 42.05 (47) | 27.67 (49)

10. Secondary Outcome: Maximum Serum Concentration (Cmax) of PF-06293620 (SAD Cohorts)
Description: Maximum serum concentration (Cmax) of PF-06293620 was observed directly from data.
Time Frame: as for outcome 4
Population: The pharmacokinetic (PK) concentration population included all enrolled participants treated who had at least 1 measurable (greater than lower limit of quantification) concentration value.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | PF-06293620 0.3 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg SC (SAD Cohorts) | PF-06293620 3.0 mg/kg SC (SAD Cohorts) | PF-06293620 6.0 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg IV (SAD Cohorts)
Number analyzed (Participants) | 6 | 5 | 6 | 7 | 6
mcg/mL | 0.3907 (58) | 2.896 (48) | 7.222 (52) | 22.30 (62) | 27.64 (20)

11. Secondary Outcome: Time for Maximum Serum Concentration (Tmax) of PF-06293620 (SAD Cohorts)
Description: Time for Maximum serum concentration (Tmax) of PF-06293620 was observed directly from data as time of first occurrence.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | PF-06293620 0.3 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg SC (SAD Cohorts) | PF-06293620 3.0 mg/kg SC (SAD Cohorts) | PF-06293620 6.0 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg IV (SAD Cohorts)
Number analyzed (Participants) | 6 | 5 | 6 | 7 | 6
hours | 168 (58) [71.9 to 336] | 168 (48) [48.0 to 504] | 252 (52) [95.9 to 504] | 168 (62) [96.0 to 504] | 1.00 (20) [1.00 to 2.00]

12. Secondary Outcome: Steady-state Volume of Distribution (Vss) of PF-06293620 (SAD Cohorts)
Description: Steady-state volume of distribution (Vss) of PF-06293620 was calculated as CL*MRT, where MRT was the mean residence time calculated as (AUMCinf/AUCinf - infusion duration/2), AUMCinf was area under the moment curve from time 0 extrapolated to infinity; CL was the clearance. This outcome measure only applies to IV arms.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | PF-06293620 1.0 mg/kg IV (SAD Cohorts)
Number analyzed (Participants) | 6
liters | 7.095 (21) [1.00 to 2.00]

13. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-06293620 (SAD Cohorts)
Description: Apparent Volume of Distribution (Vz/F) of PF-06293620 was calculated as dose/(AUCinf*kel), where AUCinf was area under the serum concentration-time profile from time 0 extrapolated to infinite time, kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. This outcome measure only applies to SC arms.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | PF-06293620 0.3 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg SC (SAD Cohorts) | PF-06293620 3.0 mg/kg SC (SAD Cohorts) | PF-06293620 6.0 mg/kg SC (SAD Cohorts)
Number analyzed (Participants) | 1 | 5 | 6 | 7
liters | 21.10 (NA) — Only 1 participant had reportable value, geometric coefficient of variation is not applicable. | 16.25 (43) | 20.63 (44) | 18.17 (48)

14. Secondary Outcome: Terminal Elimination Half-life (Thalf) of PF-06293620 (SAD Cohorts)
Description: Terminal elimination half-life (Thalf) of PF-06293620 was calculated as ln(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Only those data points judged to describe the terminal log-linear decline were used in the regression.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PF-06293620 0.3 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg SC (SAD Cohorts) | PF-06293620 3.0 mg/kg SC (SAD Cohorts) | PF-06293620 6.0 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg IV (SAD Cohorts)
Number analyzed (Participants) | 1 | 5 | 6 | 7 | 6
days | 7.33 (NA) — Only 1 participant had reportable value, geometric coefficient of variation is not applicable. | 10.95 (3.74) | 14.66 (4.21) | 19.23 (3.45) | 14.37 (3.13)

15. Secondary Outcome: Area Under the Concentration-Time Profile From Time 0 to Time Tau (AUCtau) of PF-06293620 (MAD Cohorts) After Day 1 and Day 57 Administration
Description: Tau refers to the dosing interval, which was 4 weeks (672 hours). Area under the concentration-time profile from time 0 to time tau (AUCtau) was determined using linear/log trapezoidal method.
Time Frame: Pre-dose, 1 and 4 hours post-dose on Day 1; Days 2, 3, 7, 8, 15, 27, 28; pre-dose, 1 and 4 hours post-dose on Day 29; Days 36, 43; pre-dose, 1 and 4 hours post-dose on Day 57; Days 58, 59, 63, 64, 71, 78, 84, 85, 99, 113, 141, 169
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL
Arm/Group | PF-06293620 50 mg SC (MAD Cohorts) | PF-06293620 75 mg SC (MAD Cohorts) | PF-06293620 150 mg SC (MAD Cohorts)
Number analyzed (Participants) | 8 | 16 | 8
mcg*hr/mL
  Day 1 | 609.6 (137) | 802.5 (79) | 2752 (73)
  Day 57: number analyzed (Participants) | 7 | 14 | 7
  Day 57 | 1309 (60) | 2991 (57) | 6121 (48)

16. Secondary Outcome: Maximum Serum Concentration (Cmax) of PF-06293620 (MAD Cohorts) After Day 1 and Day 57 Administration
Time Frame: as for outcome 15
Population: The PK concentration population included all enrolled participants treated who had at least 1 measurable concentration value.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | PF-06293620 50 mg SC (MAD Cohorts) | PF-06293620 75 mg SC (MAD Cohorts) | PF-06293620 150 mg SC (MAD Cohorts)
Number analyzed (Participants) | 8 | 16 | 8
mcg/mL
  Day 1 | 1.526 (139) | 1.706 (72) | 5.184 (73)
  Day 57: number analyzed (Participants) | 8 | 14 | 7
  Day 57 | 1.989 (183) | 6.012 (65) | 11.74 (56)

17. Secondary Outcome: Average Concentration (Cav) of PF-06293620 (MAD Cohorts) After Day 1 and Day 57 Administration
Description: Average Concentration (Cav) of PF-06293620 was calculated as AUCtau/tau, where AUCtau was area under the concentration-time profile from time 0 to time tau, and tau was the dosing interval, 4 weeks (672 hours).
Time Frame: as for outcome 15
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | PF-06293620 50 mg SC (MAD Cohorts) | PF-06293620 75 mg SC (MAD Cohorts) | PF-06293620 150 mg SC (MAD Cohorts)
Number analyzed (Participants) | 8 | 16 | 8
mcg/mL
  Day 1 | 0.9067 (137) | 1.194 (79) | 4.096 (73)
  Day 57: number analyzed (Participants) | 7 | 14 | 7
  Day 57 | 1.948 (60) | 4.449 (57) | 9.102 (48)

18. Secondary Outcome: Lowest Concentration Observed During the Dosing Interval (Cmin) of PF-06293620 (MAD Cohorts) After Day 57 Administration
Time Frame: Pre-dose, 1 and 4 hours post-dose on Day 57; Days 58, 59, 63, 64, 71, 78, 84, 85, 99, 113, 141, 169
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | PF-06293620 50 mg SC (MAD Cohorts) | PF-06293620 75 mg SC (MAD Cohorts) | PF-06293620 150 mg SC (MAD Cohorts)
Number analyzed (Participants) | 7 | 14 | 7
µg/mL | 0.7555 (94) | 1.979 (72) | 5.456 (48)

19. Secondary Outcome: Time for Maximum Serum Concentration (Tmax) of PF-06293620 (MAD Cohorts) After Day 1 and Day 57 Administration
Description: Time for maximum serum concentration (Tmax) of PF-06293620 was observed directly from data as time of first occurrence.
Time Frame: as for outcome 15
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | PF-06293620 50 mg SC (MAD Cohorts) | PF-06293620 75 mg SC (MAD Cohorts) | PF-06293620 150 mg SC (MAD Cohorts)
Number analyzed (Participants) | 8 | 16 | 8
hours
  Day 1 | 240 [144 to 338] | 252 [48.0 to 338] | 360 [144 to 648]
  Day 57: number analyzed (Participants) | 8 | 14 | 7
  Day 57 | 168 [47.8 to 192] | 144 [47.5 to 648] | 120 [48.0 to 504]

20. Secondary Outcome: Apparent Clearance (CL/F) of PF-06293620 (MAD Cohorts) After Day 57 Administration
Description: Apparent clearance (CL/F) of PF-06293620 was calculated as dose/AUCtau, where AUCtau was area under the concentration-time profile from time 0 to time tau, and tau was the dosing interval, 4 weeks (672 hours).
Time Frame: Pre-dose, 1 and 4 hours post-dose on Day 57; Days 58, 59, 63, 64, 71, 78, 84, 85, 99, 113, 141, 169
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr
Arm/Group | PF-06293620 50 mg SC (MAD Cohorts) | PF-06293620 75 mg SC (MAD Cohorts) | PF-06293620 150 mg SC (MAD Cohorts)
Number analyzed (Participants) | 7 | 14 | 7
mL/hr | 38.19 (60) | 25.07 (57) | 24.53 (47)

21. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-06293620 (MAD Cohorts) After Day 57 Administration
Description: Apparent volume of distribution (Vz/F) of PF-06293620 was calculated as dose/(AUCtau/kel), where AUCtau was area under the concentration-time profile from time 0 to time tau, and tau was the dosing interval, 4 weeks (672 hours); and kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Only those data points judged to describe the terminal log-linear decline were used in the regression.
Time Frame: Pre-dose, 1 and 4 hours post-dose on Day 57; Days 58, 59, 63, 64, 71, 78, 84, 85, 99, 113, 141, 169
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | PF-06293620 50 mg SC (MAD Cohorts) | PF-06293620 75 mg SC (MAD Cohorts) | PF-06293620 150 mg SC (MAD Cohorts)
Number analyzed (Participants) | 7 | 14 | 7
liters | 13.43 (38) | 10.45 (52) | 12.09 (40)

22. Secondary Outcome: Terminal Elimination Half-life (Thalf) of PF-06293620 (MAD Cohorts) After Day 57 Administration
Description: as for outcome 14
Time Frame: Pre-dose, 1 and 4 hours post-dose on Day 57; Days 58, 59, 63, 64, 71, 78, 84, 85, 99, 113, 141, 169
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PF-06293620 50 mg SC (MAD Cohorts) | PF-06293620 75 mg SC (MAD Cohorts) | PF-06293620 150 mg SC (MAD Cohorts)
Number analyzed (Participants) | 7 | 14 | 7
days | 10.37 (2.22) | 12.72 (4.21) | 14.50 (2.81)

23. Secondary Outcome: Observed Accumulation Ratio Based on AUC (Rac) of PF-06293620 (MAD Cohorts)
Description: Observed accumulation ratio based on AUC (Rac) of PF-06293620 was calculated as AUCtau(Day57)/AUCtau(Day1).
Time Frame: as for outcome 15
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06293620 50 mg SC (MAD Cohorts) | PF-06293620 75 mg SC (MAD Cohorts) | PF-06293620 150 mg SC (MAD Cohorts)
Number analyzed (Participants) | 7 | 14 | 7
ratio | 1.833 (64) | 3.446 (36) | 2.148 (30)

24. Secondary Outcome: Observed Accumulation Ratio Based on Cmax (Rac,Cmax) of PF-06293620 (MAD Cohorts)
Description: Observed accumulation ratio based on Cmax (Rac,Cmax) of PF-06293620 was calculated as Cmax(Day57)/Cmax(Day1).
Time Frame: as for outcome 15
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06293620 50 mg SC (MAD Cohorts) | PF-06293620 75 mg SC (MAD Cohorts) | PF-06293620 150 mg SC (MAD Cohorts)
Number analyzed (Participants) | 8 | 14 | 7
ratio | 1.302 (114) | 3.257 (42) | 2.188 (22)

ADVERSE EVENTS:
Time Frame: Days 1 to 85 for SAD cohorts and Days 1 to 169 for MAD cohorts; participants with positive anti-drug antibody (ADA) results were followed up to stabilization of ADA titers or up to 9 months after Day 169 visit.
Description: MedDRA 19.0 was used for SAD cohorts, and MedDRA 20.0 was used for MAD cohorts.
Arm/Group | Placebo SC (SAD Cohorts) | PF-06293620 0.3 mg/kg SC (SAD Cohorts) | PF-06293620 1.0 mg/kg SC (SAD Cohorts) | PF-06293620 3.0 mg/kg SC (SAD Cohorts) | PF-06293620 6.0 mg/kg SC (SAD Cohorts) | Placebo IV (SAD Cohorts) | PF-06293620 1.0 mg/kg IV (SAD Cohorts) | Placebo SC (MAD Cohorts) | PF-06293620 50 mg SC (MAD Cohorts) | PF-06293620 75 mg SC (MAD Cohorts) | PF-06293620 150 mg SC (MAD Cohorts)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/6 | 0/9 | 0/2 | 0/6 | 0/8 | 0/8 | 0/16 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/6 | 0/6 | 0/6 | 0/9 | 0/2 | 0/6 | 0/8 | 0/8 | 1/16 | 2/8
Other Adverse Events (participants affected / at risk) | 5/9 | 3/6 | 3/6 | 5/6 | 5/9 | 0/2 | 3/6 | 4/8 | 4/8 | 11/16 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo SC (SAD Cohorts) (N=9) | PF-06293620 0.3 mg/kg SC (SAD Cohorts) (N=6) | PF-06293620 1.0 mg/kg SC (SAD Cohorts) (N=6) | PF-06293620 3.0 mg/kg SC (SAD Cohorts) (N=6) | PF-06293620 6.0 mg/kg SC (SAD Cohorts) (N=9) | Placebo IV (SAD Cohorts) (N=2) | PF-06293620 1.0 mg/kg IV (SAD Cohorts) (N=6) | Placebo SC (MAD Cohorts) (N=8) | PF-06293620 50 mg SC (MAD Cohorts) (N=8) | PF-06293620 75 mg SC (MAD Cohorts) (N=16) | PF-06293620 150 mg SC (MAD Cohorts) (N=8)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0/8 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo SC (SAD Cohorts) (N=9) | PF-06293620 0.3 mg/kg SC (SAD Cohorts) (N=6) | PF-06293620 1.0 mg/kg SC (SAD Cohorts) (N=6) | PF-06293620 3.0 mg/kg SC (SAD Cohorts) (N=6) | PF-06293620 6.0 mg/kg SC (SAD Cohorts) (N=9) | Placebo IV (SAD Cohorts) (N=2) | PF-06293620 1.0 mg/kg IV (SAD Cohorts) (N=6) | Placebo SC (MAD Cohorts) (N=8) | PF-06293620 50 mg SC (MAD Cohorts) (N=8) | PF-06293620 75 mg SC (MAD Cohorts) (N=16) | PF-06293620 150 mg SC (MAD Cohorts) (N=8)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hunger (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site hemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Infective glossitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liver function test increased (Investigations) | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 5
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetic dermopathy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Originally planned 250 mg cohort was not enrolled in MAD part, because 150 mg cohort already demonstrated optimal glucose-lowering effect. Protocol-specified TBD (to be determined) dose level was 50 mg as well as expansion of the 75 mg cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-10-02): https://cdn.clinicaltrials.gov/large-docs/61/NCT02211261/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT02211261/SAP_001.pdf